CLINICAL TRIAL: NCT07087301
Title: A Prospective Observational Study to Analyze Factors Influencing Vancomycin Blood Concentrations in Post-Cardiac Surgery Patients Under Extracorporeal Circulation
Brief Title: Vancomycin Concentration Analysis in Post-Cardiac Surgery Patients
Status: Completed | Type: Observational
Sponsor: Pengqiang Du (Other)
Responsible Party: Sponsor-Investigator, Pengqiang Du, Associate Chief Pharmacist, Chinese Academy of Medical Sciences, Fuwai Hospital
Organization: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Other Study IDs: 2023-Ethics79
Record Dates: First submitted 2025-07-08; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2024-12

CONDITIONS: Cardiac Surgery Requiring Cardiopulmonary Bypass

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- nephrotoxicity risk group: nephrotoxicity risk group (≥20 mg/L vs <20 mg/L, n=350). A dual-model framework was established based on vancomycin's therapeutic window (10-20 mg/L): the first model (for nephrotoxicity risk prediction) defined high concentration as ≥20 mg/L and control as <20 mg/L to identify risk factors for vancomycin accumulation.
  Interventions: Other: subtherapeutic concentration risk group; Drug: subtherapeutic concentration risk group

INTERVENTIONS:
Other: subtherapeutic concentration risk group — The second model (for subtherapeutic concentration risk prediction) defined low concentration as trough <10 mg/L and target as 10-20 mg/L to analyze predictors of target concentration attainment.
Drug: subtherapeutic concentration risk group — The second model (for subtherapeutic concentration risk prediction) defined low concentration as trough <10 mg/L and target as 10-20 mg/L to analyze predictors of target concentration attainment.

SUMMARY:
The benefits of antimicrobial prophylaxis for cardiac surgery have been clearly demonstrated in placebo-controlled studies. Prophylactic intravenous antibiotics are therefore administered, with agent selection directed against the most common skin-colonising and gram-negative bacteria. Controversy persists regarding the optimal antimicrobial choice and duration of administration for cardiac surgery. In settings with a high incidence of methicillin-resistant Staphylococcus aureus (MRSA), administration of cefazolin or vancomycin for prophylaxis is considered reasonable (Class IIB recommendation, Level of Evidence C).

Vancomycin, a glycopeptide antibiotic, is widely used to treat serious gram-positive infections, including those caused by MRSA and methicillin-resistant Staphylococcus epidermidis (MRSE). Extensive pharmacokinetic/pharmacodynamic (PK/PD) studies reveal marked variability in population PK parameters across patient groups; clearance variability may reach 45 % and volume of distribution variability 48 %.

Oral vancomycin absorption is poor (≈5 % bioavailability), yet luminal concentrations remain sufficiently high for efficacy against Clostridioides difficile-associated pseudomembranous colitis. Inter-individual PK variability is substantial; two- or three-compartment models are typically employed. Protein binding ranges from 30 % to 50 %. Approximately 90 % of the dose is eliminated unchanged via the kidneys; biliary elimination is minimal. The elimination half-life is 4-7 h in individuals with normal renal function and is prolonged in patients >65 years or with renal impairment. Obesity, age, renal function, concomitant medications, disease state, and peri-operative interventions can all influence vancomycin clearance and apparent volume of distribution, potentially yielding sub- or supra-therapeutic serum concentrations.

To characterise current therapeutic drug monitoring (TDM) practices for vancomycin in cardiac-surgery patients undergoing cardiopulmonary bypass, this retrospective study combined multimodal data to develop a prognostic model predicting high- or low-risk vancomycin serum levels post-operatively. Model performance was evaluated to provide an evidence base for individualised dosing strategies aimed at optimising efficacy and minimising adverse effects.

Pharmacokinetic datasets from post-cardiac-surgery patients receiving cardiopulmonary bypass were analysed to identify determinants of vancomycin blood concentrations. Integration of baseline characteristics and medication records supports early intervention guidance for individualised vancomycin dosing and optimisation of anti-infective therapy.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing cardiac surgery with cardiopulmonary bypass
* Received intravenous vancomycin postoperatively for infection prophylaxis or treatment

Exclusion Criteria:

* Age <18 years
* Missing data on weight, height, or serum creatinine during vancomycin therapy
* No vancomycin trough plasma concentration recorded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients requiring cardiac surgery for conditions such as valvular heart disease who received postoperative vancomycin for infections.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Vancomycin trough concentration | Day 3 pre-dose
  Pre-dose vancomycin serum concentration at steady state

SECONDARY OUTCOMES:
Cardiopulmonary Bypass Duration | Intra-operative (from initiation to termination of bypass)
  Duration of cardiopulmonary bypass during cardiac surgery, recorded from initiation to termination.
Creatinine Clearance | Baseline
  Calculated using Cockcroft-Gault equation

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai Central China Cardiovascular Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No